CLINICAL TRIAL: NCT02298127
Title: Acceptability and Potential Efficacy of a Randomised, Double-blinded, Sham-controlled Trial of Auricular Acupressure for Smoking Cessation: A Pilot Study
Brief Title: Auricular Acupressure for Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Yim Wah Mak, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AASC101114
Record Dates: First submitted 2014-11-16; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; auricular acupressure; primary care settings; randomized controlled trial
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Shenmen, mouth, lung & stomach (Experimental): Participants in this group will receive 4 weekly treatment sessions of auricular acupressure via the shenmen, mouth, lung and stomach.
  Interventions: Other: Auricular acupressure
- Subcortex,endocrine&sympathetic systems (Experimental): Participants in this group will receive 4 weekly treatment sessions of auricular acupressure via the subcortex, endocrine and sympathetic systems.
  Interventions: Other: Auricular acupressure
- Elbow, shoulder & knee (Sham Comparator): Participants in this group will receive 4 weekly treatment sessions of sham-controlled acupressure on the elbow, shoulder and knee acupoints on the auricle that is non-specific to smoking cessation.
  Interventions: Other: Auricular acupressure

INTERVENTIONS:
Other: Auricular acupressure — For each auricular acupressure weekly session, magnetic ears tacks will be will be applied by certified traditional Chinese medicine practitioners according to the allocated group assignment, for a duration of one month.

SUMMARY:
The purpose of this study is to evaluate the potential efficacy of auricular acupressure to stimulate specific acupoints in enhancing smoking cessation by reducing nicotine withdrawal symptoms among attendees in primary healthcare settings.

DETAILED DESCRIPTION:
Uncontrolled trials indicated that auricular acupressure is an effective treatment for addictive behaviors such as smoking cessation. However, some methodological limitations can be identified among clinical trials in this area, and it is not clear whether it is more efficacious to use the commonly-used acupoints or other points that are specifically for reducing the withdrawal symptoms of nicotine. The study addresses the identified methodological shortcomings of the previous similar studies. It consists of a total of three intervention groups, which allows comparisons between the commonly-used acupoints of acupressure, acupoints specific to smoking cessation, and a sham-controlled intervention. The study does not only focus on the efficacy of smoking cessation but also assesses the mediate effect of auricular acupressure on nicotine withdrawal by questionnaire and biomarkers.

This is the first study of its kind to yield information on the acceptability and effectiveness of a safe, available auricular acupressure technique on smoking cessation in Hong Kong. The findings could provide further information for the development of future tobacco-control activities targeting smokers in a wider population who would like to use acupressure as a treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Currently smoking at least one cigarette per day in the past 30 days
* Are Hong Kong residents
* Able to communicate in Cantonese
* Currently reside in Hong Kong and expect to continue to do so for the next 6 months
* Have access to a telephone

Exclusion Criteria:

* Currently undergoing other smoking cessation or similar programme
* With a known history of allergy to adhesive tapes or history of current otitis externa or other ear disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence by self report | 1.25 month after the initial contact
7-day point prevalence by self report, validated by biochemical measures | 6 month
  Obtaining CO measurement and testing urinary cotinine for those participants who report quitting smoking
Withdrawal symptoms | 1.25 month after the initial contact
  Measured by two biomarkers for nicotine dependence: the gene expression level of nicotinic acetylcholine receptors (nAChRs) and dopamine level

SECONDARY OUTCOMES:
Feasibility outcome assessed in terms of participant recruitment, acupressure session attendance, retention, preference for using TCM for smoking cessation, perceived usefulness and confidence of quitting smoking by acupressure | 6 month
  Feasibility outcomes will be assessed in terms of participant recruitment, acupressure session attendance, retention, preference for using TCM for smoking cessation, perceived usefulness and confidence of quitting smoking by acupressure
Acceptability: Subjective data on acceptability of auricular acupressure for smoking cessation | 1 month
  Subjective data on acceptability of auricular acupressure for smoking cessation will be collected at each visit

CONTACTS AND LOCATIONS:
Overall Officials: YW Mak, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong